CLINICAL TRIAL: NCT00624273
Title: Effect of Sildenafil on Digital Ulcers in Systemic Sclerosis
Brief Title: Sildenafil for Treatment of Digital Ulcers in Patients With Systemic Sclerosis
Acronym: Sildenafil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: PD Dr. Gabriela Riemekasten, Charité Universitäsmedizin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDN-D-002G; SDN-D-002G
Record Dates: First submitted 2008-02-14; First posted 2008-02-27 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2003-07

CONDITIONS: Active Digital Ulcers
Keywords: digital ulcers,; systemic sclerosis,; sildenafil,; vasoactive therapies
MeSH Terms: conditions — digital ulcers; Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1, active ulcers (Other): sildenafil treatment
  Interventions: Drug: Sildenafil therapy

INTERVENTIONS:
Drug: Sildenafil therapy — oral use
  Other Names: start at 25 mg

SUMMARY:
This is a pilot study analyzing the effect of sildenafil therapy on digital ulcers in systemic sclerosis. We want to analyze ulcer healing by measuring the size of digital ulcers and their count and analyze the effect of sildenafil on angiography.

DETAILED DESCRIPTION:
INVESTIGATOR: Dr. Gabriela Riemekasten Anke Praast Prof. G. R. Burmester Prof. Falk Hiepe

OBJECTIVES:

Sildenafil is a very potent drug in the treatment of digital ulcers secondary to Raynaud´s phenomenon in patients with connective tissue diseases. Probably, sildenafil has a disease-modifying capability improving different signs of a disturbed regulation of vascular tone in connective tissue diseases. Sildenafil can be used over a long period without significant side effects in scleroderma patients and improves disease severity, life quality, and prognosis of patients with connective tissue diseases and secondary Raynaud's phenomenon.

SUBJECTS and CENTERS:

We want to study 10-15 patients with digital ulcers secondary to connective tissue diseases and which are refractory to other drugs, such as calcium channel blockers or iloprost. In this pilot study, patients are treated only in the Charité University Hospital.

INCLUSION/EXCLUSION CRITERIA

1 . Digital gangrene, ulcers in patients with severe secondary Raynaud's phenomenon

2. Stable therapy with vasoactive drugs, such as calcium channel blockers, angiotensin inhibitors/AT II receptor antagonists or pentoxifyllin 4 weeks before and during the treatment with sildenafil.

3. Unchanged immunosuppressive therapy 3 months before treatment with sildenafil

4. No effect of prostacyclin treatment, contraindications for prostacyclins, or other reasons excluding this therapy

EXCLUSION CRITERIA:

1. Therapy with iloprost during the last 4 weeks
2. Sympathectomy during the last 4 weeks
3. TIA, stroke, myocardial infarction during the last 6 months
4. Instable angina pectoris
5. Hemorrhagic diathesis, thrombocytic dysfunction, fibromuscular dysplasia
6. Microangiopathic hemolytic anaemia
7. Azotaemia
8. Hypertonus not adjustable with diuretic, clonidine, ACE inhibitors/AT II antagonists, calcium channel blockers)
9. Left ventricular ejection fraction< 20%
10. Hypotonus < 80/40 mm Hg
11. Positive pregnancy test
12. History of cancer
13. History of gastric/duodenic ulcers without endoscopic proof of complete healing
14. Participation in other studies (currently or during the last 4 weeks)
15. Abuse of alcohol or other drugs, smoker
16. Cardiac failure, use of nitrates

STUDY DESIGN:

This is an open prospective pilot study of one centre determining the effect of a 6 month treatment of sildenafil in patients with acral ulcers in secondary Raynaud's phenomenon due to connective tissue diseases.

Drop out criteria's/ final points:

1 . Any change of the immunomodulating or suppressing therapy (e.g., treatment with cyclophosphamide because of an alveolitis; bolus of steroids > 30 mg/d).

2. No response on the healing of ulcers after 4 weeks of treatment with sildenafil 3. Manifestation of new ulcers/necrosis under sildenafil 4. Escalation of medication with an vascular influence (calcium channel blockers, ACE inhibitors/AT II receptor blockers)

ELIGIBILITY:
Inclusion Criteria:

1. Digital gangrene, ulcers in patients with severe secondary Raynaud's phenomenon
2. Stable therapy with vasoactive drugs, such as calcium channel blockers, angiotensin inhibitors/AT II receptor antagonists or pentoxifyllin 4 weeks before and during the treatment with sildenafil.
3. Unchanged immunosuppressive therapy 3 months before treatment with sildenafil
4. No effect of prostacyclin treatment, contraindications for prostacyclins, or other reasons excluding this therapy

Exclusion Criteria:

1. Therapy with iloprost during the last 4 weeks
2. Sympathectomy during the last 4 weeks
3. TIA, stroke, myocardial infarction during the last 6 months
4. Instable angina pectoris
5. Hemorrhagic diathesis, thrombocytic dysfunction, fibromuscular dysplasia
6. Microangiopathic hemolytic anaemia
7. Azotaemia
8. Hypertonus not adjustable with diuretic, clonidine, ACE inhibitors/AT II antagonists, calcium channel blockers)
9. Left ventricular ejection fraction< 20%
10. Hypotonus < 80/40 mm Hg
11. Positive pregnancy test
12. History of cancer
13. History of gastric/duodenic ulcers without endoscopic proof of complete healing
14. Participation in other studies (currently or during the last 4 weeks)
15. Abuse of alcohol or other drugs, smoker
16. Cardiac failure, use of nitrates

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-02; Primary Completion 2004-11 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
healing of digital ulcer | 6 months

SECONDARY OUTCOMES:
Decrease of frequency/duration of Raynaud's attacks (monthly) | 6 months
Prevention of necroses manifestations | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gabriela Riemekasten, MD, Principal Investigator — Charité Universitätsklinik Berlin
Locations (1):
- Riemekasten, PD Dr. med., Berlin, State of Berlin, Germany